CLINICAL TRIAL: NCT00861029
Title: A Randomized, Blinded Placebo-Controlled Study to Evaluate the Effect of Repeat Oral Doses of Pazopanib (GW786034) on the Electrocardiogram (ECG) With Focus on Cardiac Repolarization (QTc Duration) in Subjects With Solid Tumors
Brief Title: VEG111485: A QTc Study of Pazopanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111485
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: GW786034, pazopanib, moxifloxacin, ECG intervals and morphology, QTc, Holter monitor, pharmacokinetics, safety, cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — pazopanib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazopanib (Experimental): Subjects will receive pazopanib during study
  Interventions: Drug: Pazopanib; Drug: Moxifloxacin; Other: Placebo for moxifloxacin
- Placebo (Other): Placebo as a comparator to pazopanib
  Interventions: Other: Placebo for pazopanib; Drug: Moxifloxacin; Other: Placebo for moxifloxacin

INTERVENTIONS:
Drug: Pazopanib — Subjects treated with pazopanib
  Arms: Pazopanib
Other: Placebo for pazopanib — Control for comparison with pazopanib
  Arms: Placebo
Drug: Moxifloxacin — Comparator for pazopanib
Other: Placebo for moxifloxacin — Placebo for moxifloxacin

SUMMARY:
This is a Phase I, randomized, double-blind, placebo-controlled, study to estimate the effects of daily oral dosing of 800 mg pazopanib on electrocardiographic parameters (QTc interval duration) as compared with placebo in subjects with solid tumors. Moxifloxacin, will serve as a positive control.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo-controlled, parallel group study designed to estimate the effects of repeated, once daily oral dosing of pazopanib on electrocardiographic parameters with a particular focus on its effect on cardiac repolarization (QTc interval duration) as compared with placebo in subjects with solid tumors. Moxifloxacin, a drug known to cause mild QTc interval prolongation, is included as a positive control to validate the ability of the study to detect a small prolongation in the QTc interval. Digital 12-lead electrocardiograms (ECGs) will be extracted from continuous ECG recordings obtained via a Holter monitor. The effects of pazopanib and moxifloxacin on cardiac repolarization will be compared with placebo.

This study will also assess the pharmacokinetic-pharmacodynamic relationship between plasma concentrations of pazopanib and its metabolites and their effects, if any, on cardiac repolarization, specifically on the QT interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older, at the time of signing of the informed consent.
* Has histologically or cytologically confirmed advanced solid tumor malignancy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Able to swallow and retain oral medication.
* Adequate organ systems function.
* Serum potassium level >4 mEq/L, magnesium level >1.7 mg/dL and total serum calcium level within normal limits (if albumin is <4.5 g/dL, albumin-corrected total serum calcium level should be within normal limits [see Appendix 7]). NOTE: Supplementation is permitted in order to meet this criterion. Subject should be retested following supplementation.
* Subject is a woman of non-childbearing potential or willing to use acceptable contraception.
* Subject is a man with a female partner of childbearing potential agrees to use contraception.
* Subject, if sexually active, agrees to continue the recommended contraception method for the duration of treatment and for 28 days following discontinuation of treatment.
* Capable of giving written informed consent.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any of the following ECG findings, QTcF interval >470 msec, PR interval >240 msec or ≤110msec, Bradycardia defined as sinus rate <50 beats per minute
* Cardiac conduction abnormalities denoted by any of the following: Evidence of second-degree (type II) or third-degree atrioventricular block, Evidence of ventricular pre-excitation, Electrocardiographic evidence of complete left bundle branch block (LBBB), Intraventricular conduction delay with QRS duration >120 msec, Atrial fibrillation, Presence of cardiac pacemaker.
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, symptomatic peripheral vascular disease or other clinically significant cardiac disease.
* For subjects with a history of myocardial infarction (>6 months ago), congestive heart failure (>6 months ago) or prior anthracycline exposure, left ventricular ejection fraction (LVEF) must be assessed within 28 days prior to the first dose of study drug by one of the following methods: multiple gated acquisition (MUGA) scan or echocardiogram (ECHO). Subjects with a measurement of LVEF <50% are excluded from participation in the study.
* Personal or family history of long-QT syndrome.
* History or clinical evidence of CNS metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 2 months prior to beginning study treatment.
* Clinically significant gastrointestinal (GI) abnormalities that may affect the absorption of study drug including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel.
* Clinically significant GI abnormalities that may increase the risk for GI bleeding including, but not limited to: active peptic ulcer disease, known intra-luminal metastatic lesion(s) with suspected bleeding, inflammatory bowel disease, ulcerative colitis or other GI conditions with increased risk of perforation, history of abdominal fistula, GI perforation or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Presence of uncontrolled infection.
* Unable or unwilling to discontinue use of prohibited medications listed in Section 9.2 for at least 14 days prior to the first dose of study drug (see Section 9.2).
* Poorly controlled hypertension [systolic blood pressure (SBP) >140 mmHg, or diastolic blood pressure (DBP) >90 mmHg].
* History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Evidence of active bleeding or bleeding diathesis.
* Hemoptysis within 6 weeks prior to the first dose of study drug.
* Known endobronchial lesion(s) or involvement of large pulmonary vessel(s) by tumor.
* History of sensitivity or allergic reaction to moxifloxacin or any member of the quinolone class of antimicrobial agents.
* Treatment with anti-cancer therapy (including chemotherapy, radiation therapy, immunotherapy, biologic therapy, investigational therapy, hormonal therapy, surgery or tumor embolization) within 14 days prior to the first dose of pazopanib.
* History or presence of hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Prior major surgery or trauma within the past 28 days prior to the first dose of study drug and/or presence of any non-healing wound, fracture or ulcer.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03-19 (Actual); Primary Completion 2010-02-15 (Actual); Study Completion 2010-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF interval at each time point on Study Day 9 (average of at least 3 Holter ECG replicates per time point) as compared with time-matched placebo. | 11 days

SECONDARY OUTCOMES:
ECG parameters: RR interval, QT, QTcB, heart rate, PR, QRS intervals and morphology. | 11 days
Plasma pazopanib and metabolites (GSK1268992, GSK1268997 and GSK1071306) concentrations and PK parameters AUC(0-t), AUC(0-24), C24 Cmax and tmax as data permit. | 11 days
Change from baseline in QTcF interval at each time point on Study Day 1 (average of at least 3 Holter ECG replicates per time point) as compared with time-matched placebo. | 11 days
Plasma moxifloxacin concentrations and PK parameters AUC(0-t), AUC(0-∞), Cmax and tmax as data permit. | 11 days
Safety parameters: AEs, vital signs, ECGs and clinical laboratory assessments. | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tacoma, Washington

REFERENCES:
- [Background] Heath EI, Infante J, Lewis LD, Luu T, Stephenson J, Tan AR, Kasubhai S, LoRusso P, Ma B, Suttle AB, Kleha JF, Ball HA, Dar MM. A randomized, double-blind, placebo-controlled study to evaluate the effect of repeated oral doses of pazopanib on cardiac conduction in patients with solid tumors. Cancer Chemother Pharmacol. 2013 Mar;71(3):565-73. doi: 10.1007/s00280-012-2030-8. Epub 2013 Jan 24. PMID 23344712
- See also: Results for study 111485 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111485?search=study&study_ids=111485#rs